CLINICAL TRIAL: NCT01348139
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Multicentre, 6-way Crossover, Single-dose, Phase IIa Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Different Dry Powder Inhalation Formulations of AZD3199 Administered Via Single Inhalation Device Compared to AZD3199 Administered Via Turbuhaler™ Inhaler in Patients With Asthma
Brief Title: Evaluation of the Pharmacokinetics and the Pharmacodynamics of Different Dry Powder Inhalation Formulations of AZD3199 in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D0570C00011; 2011-000133-37 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
Keywords: Asthma; patients; lung function
MeSH Terms: conditions — Asthma | interventions — AZD-3199

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- 1 (Experimental): AZD3199 800 µg inhaled via single inhaler device (SID), single dose
  Interventions: Drug: AZD3199
- 2 (Experimental): AZD3199 880 µg inhaled via SID, single dose
  Interventions: Drug: AZD3199
- 3 (Experimental): AZD3199 1400 µg inhaled via SID, single dose
  Interventions: Drug: AZD3199
- 4 (Experimental): AZD3199 300 µg inhaled via Turbuhaler inhaler, single dose
  Interventions: Drug: AZD3199
- 5 (Experimental): AZD3199 1200 µg inhaled via Turbuhaler inhaler, single dose
  Interventions: Drug: AZD3199
- 6 (Placebo Comparator): Placebo inhaled via Turbuhaler inhaler and SID, single dose
  Interventions: Other: AZD3199 Placebo

INTERVENTIONS:
Drug: AZD3199 — Inhaled via single inhaler device (SID)
  Arms: 1; 2; 3
Drug: AZD3199 — Inhaled via Turbuhaler inhaler
  Arms: 4; 5
Other: AZD3199 Placebo — Inhaled via Turbuhaler inhaler and SID
  Arms: 6

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and pharmacodynamics of single doses of three different dry powder inhalation formulations of AZD3199 administered via Single Inhalation Device (SID) compared to AZD3199 administered via Turbuhaler™ Inhaler and compared to placebo in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures
* Men or women, age ≥ 18 years. Women must be of non-childbearing potential or stable on a highly effective contraceptive method for at least 3 months prior to Visit 1 and be willing to continue on the chosen contraceptive method throughout the study.
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to study start
* A history of asthma for at least 6 months.
* Body Mass Index (BMI) 19-30 kg/m2

Exclusion Criteria:

* Significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the result of the study, or the patient's ability to participate in the study
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to β2-agonists in general or to AZD3199 and/or excipients
* Prolonged QTcF > 450 msec or shortened QTcF <340 msec
* History of alcohol/drug abuse or excessive intake of alcohol as judged by the Investigator
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Lund

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 patients were enrolled at 3 centres in Sweden. Of these, 26 patients were randomised to receive a treatment sequence consisting of 6 different treatments in random order. The number of patients randomised was well balanced across all the treatment periods. In total, 25 patients completed the study.
Groups:
- 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg: AZD3199 1400 μg SID followed by Placebo followed by AZD3199 880 μg SID followed by AZD3199 1200 μg Turbuhaler inhaler followed by AZD3199 800 μg SID followed by AZD3199 300 μg Turbuhaler inhaler.
- 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg: AZD3199 880 μg SID followed by AZD3199 1400 μg SID followed by AZD3199 800 μg SID followed by Placebo followed by AZD3199 300 μg Turbuhaler inhaler followed by AZD3199 1200 μg Turbuhaler inhaler.
- 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo: AZD3199 800 μg SID followed by AZD3199 880 μg SID followed by AZD3199 300 μg Turbuhaler inhaler followed by AZD3199 1400 μg SID followed by AZD3199 1200 μg Turbuhaler inhaler followed by Placebo.
- 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg: AZD3199 300 μg Turbuhaler inhaler followed by AZD3199 800 μg SID followed by AZD3199 1200 μg Turbuhaler inhaler followed by AZD3199 880 μg SID followed by Placebo followed by AZD3199 1400 μg SID.
- 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg: AZD3199 1200 μg Turbuhaler inhaler followed by AZD3199 300 μg Turbuhaler inhaler followed by Placebo followed by AZD3199 800 μg SID followed by AZD3199 1400 μg SID followed by AZD3199 880 μg SID.
- Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg: Placebo followed by AZD3199 1200 μg Turbuhaler inhaler followed by AZD3199 1400 μg SID followed by AZD3199 300 μg Turbuhaler inhaler followed by AZD3199 880 μg SID followed by AZD3199 800 μg SID.
Period: Period 1
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 5 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 4 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 4 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 4 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 4 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | 1400 μg / Placebo / 880 μg / 1200 μg / 800 μg / 300 μg | 880 μg / 1400 μg / 800 μg / Placebo / 300 μg / 1200 μg | 800 μg / 880 μg / 300 μg / 1400 μg / 1200 μg / Placebo | 300 μg / 800 μg / 1200 μg / 880 μg / Placebo / 1400 μg | 1200 μg / 300 μg / Placebo / 800 μg / 1400 μg / 880 μg | Placebo / 1200 μg / 1400 μg / 300 μg / 880 μg / 800 μg
Started | 4 | 4 | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Total: Total number of patients randomised and treated in the study.
Arm/Group | Baseline Total
Number analyzed (Participants) | 26
Age Continuous [Mean (Standard Deviation); unit: Years]
  All | 36.5 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 24
  Asian | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Emax: Maximum Value of FEV1 for Every Treatment Visits
Description: Peak effect (Emax) within 0-24 hours of FEV1, for treatment visits 2 to 7.
Time Frame: 0-24 hrs
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Arm 1 - AZD3199 1400 μg: AZD3199 1400 μg SID
- Arm 2 - AZD3199 880 μg: AZD3199 880 μg SID
- Arm 3 - AZD3199 800 μg: AZD3199 800 μg SID
- Arm 4 - AZD3199 300 μg: AZD3199 300 μg Turbuhaler inhaler
- Arm 5 - AZD3199 1200 μg: AZD3199 1200 μg Turbuhaler inhaler
- Arm 6 - Placebo: Placebo
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Liters | 3.788 (0.782) | 3.784 (0.724) | 3.756 (0.733) | 3.763 (0.744) | 3.847 (0.781) | 3.498 (0.676)

2. Primary Outcome: E22-26h: The Average of the FEV1 Values Between 22 and 26 h for Every Treatment Visit
Description: Trough effect (E22-26h) will be computed from the repeated measurements collected after each single dose during 22-26 hours of FEV1 from visit 2 to 7.
Time Frame: 22-26 hrs.
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Liters | 3.448 (0.709) | 3.453 (0.739) | 3.495 (0.730) | 3.448 (0.732) | 3.569 (0.761) | 3.310 (0.723)

3. Secondary Outcome: tEmax: Time to Maximum Value of FEV1 for Every Treatment Visit
Description: Time to peak effect (tEmax), within 0-24 hours of FEV1, for treatment visits 2 to 7.
Time Frame: 0 - 24 hrs.
Population: PD analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Hours | 2.000 [0.50 to 10.00] | 2.000 [0.50 to 22.00] | 2.000 [0.25 to 24.00] | 1.000 [0.25 to 22.00] | 4.000 [0.25 to 24.00] | 10.000 [0.00 to 24.00]

4. Secondary Outcome: E5min: The Value of FEV1 at 5 Min for Every Treatment Visit.
Description: Onset of effect (E5min), observed at 5 min. FEV1 for treatment visits 2 to 7.
Time Frame: FEV1 at 5 min
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Liters | 3.406 (0.743) | 3.449 (0.663) | 3.496 (0.692) | 3.489 (0.653) | 3.486 (0.723) | 3.188 (0.586)

5. Secondary Outcome: E0-24h: The Average of the FEV1 Values Between 0 and 24 h for Every Treatment Visit
Description: Average effect over 0-24 hours of FEV1 (E0-24h), for treatment visits 2 to 7.
Time Frame: 0 - 24 hrs
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Liters | 3.489 (0.710) | 3.526 (0.737) | 3.537 (0.729) | 3.493 (0.707) | 3.636 (0.776) | 3.287 (0.671)

6. Secondary Outcome: Emax: Maximum Value of Pulse for Every Treatment Visits
Description: Peak effect (Emax) within 0-4 hours of pulse, for treatment visits 2 to 7.
Time Frame: 0 - 4 hrs.
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 25 | 25
Beats/min | 66.15 (11.10) | 64.36 (10.10) | 64.24 (9.27) | 64.84 (10.18) | 66.20 (12.38) | 64.12 (11.22)

7. Secondary Outcome: E0-4h: The Average of the Pulse Values Between 0 and 4 h for Every Treatment Visit
Description: Average effect (E0-4h) of Pulse, for treatment visits 2 to 7.
Time Frame: 0 - 4 hrs.
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 25 | 25
Beats/min | 59.85 (9.13) | 59.13 (8.83) | 59.07 (8.38) | 58.77 (8.66) | 59.73 (9.63) | 58.66 (10.40)

8. Secondary Outcome: Cmax: Maximum Plasma Concentration
Description: Maximum plasma concentration (Cmax) for AZD3199 doses
Time Frame: 0 - 120 hrs for first two treatment visit 2 and 3 and 0 - 48 hrs for other treatment visits.
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 25 | 0
nmol/L | 6.93846 (2.497151) | 5.81240 (2.497151) | 6.29560 (2.827910) | 3.01836 (1.294151) | 13.54120 (4.337208) |

9. Secondary Outcome: AUC: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC),
Description: Area under the plasma concentration-time curve from zero to infinity (AUC), for AZD3199 doses
Time Frame: 0 - 120 hrs for first two treatment visit 2 and 3 and 0 - 48 hrs for other treatment visits.
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 25 | 0
nmol*h/L | 21.83501 (10.43729) | 20.21716 (10.19966) | 22.80110 (11.71379) | 10.25880 (4.886541) | 37.48982 (13.11484) |

10. Secondary Outcome: Tmax:Time to Maximum Plasma Concentration
Description: Time to maximum plasma concentration (tmax), for AZD3199 doses
Time Frame: 0 - 120 hrs for first two treatment visit 2 and 3 and 0 - 48 hrs for other treatment visits.
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 25 | 0
Hours | 0.47000 [0.2300 to 0.6200] | 0.48000 [0.2700 to 0.6200] | 0.52000 [0.2800 to 1.0300] | 0.52000 [0.2500 to 0.5800] | 0.48000 [0.2700 to 0.5800] |

11. Secondary Outcome: t1/2 :Terminal Half-life
Description: Terminal half-life (t1/2),for AZD3199 doses
Time Frame: 0 - 120 hrs for first two treatment visit 2 and 3 and 0 - 48 hrs for other treatment visits.
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Arm 1 - AZD3199 1400 μg | Arm 2 - AZD3199 880 μg | Arm 3 - AZD3199 800 μg | Arm 4 - AZD3199 300 μg | Arm 5 - AZD3199 1200 μg | Arm 6 - Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 9 | 0
Hours | 80.97301 (24.65131) | 79.24210 (22.07879) | 103.7279 (113.8432) | 77.46496 (47.17895) | 88.99700 (46.23237) |

ADVERSE EVENTS:
Groups:
- AZD3199 1400 μg: AZD3199 1400 μg SID
- AZD3199 880 μg: AZD3199 880 μg SID
- AZD3199 800 μg: AZD3199 800 μg SID
- AZD3199 300 μg: AZD3199 300 μg Turbuhaler inhaler
- AZD3199 1200 μg: AZD3199 1200 μg Turbuhaler inhaler
- Placebo: Placebo
Arm/Group | AZD3199 1400 μg | AZD3199 880 μg | AZD3199 800 μg | AZD3199 300 μg | AZD3199 1200 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 9/26 | 9/25 | 7/25 | 7/25 | 14/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3199 1400 μg (N=26) | AZD3199 880 μg (N=25) | AZD3199 800 μg (N=25) | AZD3199 300 μg (N=25) | AZD3199 1200 μg (N=25) | Placebo (N=25)
VOMITING (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 5 | 0 | 3 | 3 | 5 | 4
DYSGEUSIA (Nervous system disorders) | 4 | 5 | 6 | 4 | 6 | 0
HEADACHE (Nervous system disorders) | 2 | 3 | 2 | 0 | 4 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less